CLINICAL TRIAL: NCT03667352
Title: Efficacy Of Scalp Block And Ultrasound Guided TAP Block With Clonidine As Adjuvant To Ropivacaine Versus Intravenous Fentanyl On Intraoperative Hemodynamics And Perioperative Analgesia In Abdominal Bone Flap Cranioplasties: A Prospective, Randomised, Double Blind Study
Brief Title: Efficacy Of Scalp Block And Ultrasound Guided TAP Block With Clonidine As Adjuvant To Ropivacaine Versus Intravenous Fentanyl On Intraoperative Hemodynamics And Perioperative Analgesia In Abdominal Bone Flap Cranioplasties
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dhritiman Chakrabarti (Other)
Responsible Party: Sponsor-Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Organization: National Institute of Mental Health and Neuro Sciences, India (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DNBT-61/2017
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Condition: Abdominal Bone Flap Cranioplasty; Focus of Study: Perioperative Analgesia
Keywords: Scalp block; Transversus abdominis plane block; Ropivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalp & TAP Block (Group T) (Experimental): Group T received 0.2% Ropivacaine + clonidine 1µg/kg mixture, for ipsilateral scalp block (10ml),TAP block under USG guidance (20ml) and intravenous saline 0.1ml/kg/hr (sham infusion) for continuous infusion.
  Interventions: Procedure: Unilateral Scalp Block; Procedure: Transversus abdominis plane block
- Intravenous Fentanyl (Group C) (Active Comparator): Group C received saline, for ipsilateral scalp block (10ml) and TAP block under USG guidance (20ml) and I.V fentanyl 1 µg/kg/hr as analgesic.
  Interventions: Drug: Intravenous Fentanyl

INTERVENTIONS:
Procedure: Unilateral Scalp Block — Scalp block is provided by injecting local anaesthetic in the scalp at specific areas to block 6 nerves which are responsible for sensory innervation of the scalp - Supraorbital and supratrochlear nerves, Zygomaticotemporal nerve, Auriculotemporal nerve, Greater and lesser occipital nerves.
  Arms: Scalp & TAP Block (Group T)
Procedure: Transversus abdominis plane block — The transverse abdominis plane (TAP) block is a peripheral nerve block designed to anesthetize the nerves supplying the anterior abdominal wall (T6 to L1). It is usually accomplished by a single bolus injection into the transversus abdominis plane through the lumbar triangle of Petit and can be accomplished either by blind landmark based technique or alternatively under ultrasound guidance (as in this study).
  Other Names: TAP block
  Arms: Scalp & TAP Block (Group T)
Drug: Intravenous Fentanyl — Fentanyl is a commonly used opioid drug administered for analgesia in the perioperative period. It may be used as either intermittent bolus administration or continuous infusion or a combination of the two. Usual infusion doses range from 1-2 microgram/kg/hr, which may be titrated based on intraoperative haemodynamics or postoperative patient reported pain scores.
  Arms: Intravenous Fentanyl (Group C)

SUMMARY:
This study assesses efficacy of scalp block and Ultrasound guided transverse abdominis plane (TAP) block with 1µg/kg clonidine as adjuvant to 0.2% ropivacaine versus intravenous fentanyl (0.1µg/kg/hr) on intraoperative hemodynamics and perioperative analgesia in abdominal bone flap cranioplasties (ABFC).

DETAILED DESCRIPTION:
Scalp blocks with local anaesthetic agents along with general anaesthesia provides intraoperative and postoperative analgesia by blunting the hemodynamic responses to noxious stimuli. The transversus abdominis plane "TAP" block, a regional anaesthesia technique that provides analgesia following abdominal surgery. It involves a single large bolus injection of local anaesthetic into an anatomical space between the internal oblique and transversus abdominis muscles.

Ropivacaine is less cardio toxic, less arrhythmogenic, less toxic to central nervous system (CNS) than bupivacaine, and it also has intrinsic vasoconstrictor property. Clonidine is an alpha-2 receptor agonist, which has a known property of reducing requirement of analgesics in the perioperative period.

This study aimed to assess the efficacy of scalp block and TAP block with 1µg/kg clonidine as adjuvant to 0.2% ropivacaine versus intravenous fentanyl (0.1µg/kg/hr) on intraoperative hemodynamics and perioperative analgesia in abdominal bone flap cranioplasties.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing Abdominal bone flap replacement.

Exclusion Criteria:

1. Motor and comprehensive aphasia,
2. Disoriented mental state or Inability to follow commands.
3. Hypersensitivity to amide local anesthetics,
4. Bone flap site infection
5. Coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Difference in Postoperative Rescue Analgesia requirement between groups | Measured at 1, 6 and 24 hours postoperatively.
  Postoperative rescue analgesia (Inj. paracetamol 1gm I.V) if patient reported pain measured by visual analogue score was ≥ 4.
  Visual analogue scale (VAS) is a self reported score for estimation of pain which ranges between 1 (no pain) to 10 (worst possible pain).
  VAS score interpretation: No pain - 1, Mild pain <4, Moderate pain 4-7, Severe pain >7, Worst possible pain =10.

SECONDARY OUTCOMES:
Difference in intraoperative trend of Heart rate between groups | Measured at 10, 20, 30, 40, 50, 60, 90, 120, 150, 180 minutes after anaesthesia induction.
  Heart rate measured intraoperatively will be compared between the groups.
Difference in intraoperative trend of Systolic blood pressure between groups | Measured at 10, 20, 30, 40, 50, 60, 90, 120, 150, 180 minutes after anaesthesia induction.
  Systolic blood pressure measured intraoperatively will be compared between the groups.
Difference in intraoperative trend of Diastolic blood pressure between groups | Measured at 10, 20, 30, 40, 50, 60, 90, 120, 150, 180 minutes after anaesthesia induction.
  Diastolic blood pressure measured intraoperatively will be compared between the groups.
Difference in patient reported postoperative pain | Measured at 1, 6 and 24 hours postoperatively.
  Postoperative pain measured by measured by visual analogue scoring system (VAS).
  Range: 1-10. No pain - 1, Mild pain <4, Moderate pain 4-7, Severe pain >7, Worst possible pain =10.

CONTACTS AND LOCATIONS:
Locations (1):
- Yashoda Hospitals, Secunderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No